CLINICAL TRIAL: NCT01219075
Title: Soy Treatment for High-risk Women
Brief Title: Soy Isoflavones Supplementation in Treating Women at High Risk For or With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); California Breast Cancer Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1B-10-6; NCI-2010-01847
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Soybean Proteins; Magnetic Resonance Spectroscopy; Biopsy; Immunohistochemistry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral soy isoflavones supplement once daily for 12 months in the absence of disease progression.
  Interventions: Dietary Supplement: soy isoflavones; Other: questionnaire administration; Procedure: magnetic resonance imaging; Procedure: biopsy; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: mammography
- Arm II (Placebo Comparator): Patients receive oral placebo once daily for 12 months in the absence of disease progression.
  Interventions: Other: placebo; Other: questionnaire administration; Procedure: magnetic resonance imaging; Procedure: biopsy; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: mammography

INTERVENTIONS:
Dietary Supplement: soy isoflavones — Given orally
  Other Names: NovaSoy; soy phytoestrogens
  Arms: Arm I
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II
Other: questionnaire administration — Ancillary studies
Procedure: magnetic resonance imaging — Correlative studies
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Other: laboratory biomarker analysis — Correlative studies
Procedure: mammography — Correlative studies

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of soy isoflavones supplements may prevent or treat early stage breast cancer. PURPOSE: This clinical trial studies soy isoflavones supplementation in treating women at high risk for or with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess whether magnetic resonance imaging (MRI) volume (equivalent to 3-dimensional mammographic density) is reduced in high-risk women or those with invasive breast cancer or DCIS who are supplemented daily with soy (5p mg total isoflavones as aglycone) compared to placebo (microcrystalline cellulose) tablets for 1 year.II. To assess whether cell proliferation and apoptosis, as measured by Ki67 and caspase 3 staining, respectively, of breast epithelial cells is altered with soy treatment.SECONDARY OBJECTIVES: I. To assess whether other intermediate molecular markers including estrogen receptor alpha (ER alpha) and ER beta differ between women supplemented with soy vs placebo. OUTLINE: Patients are randomized to 1 of 2 treatment arms.ARM I: Patients receive oral soy isoflavones supplement once daily for12 months in the absence of disease progression.ARM II: Patients receive oral placebo once daily for 12 months in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Women at high risk for breast cancer, defined as any of the following groups:
* Five year Gail risk > 1.7%
* Known BRCA1/BRCA2 mutation carrier
* Family history consistent with hereditary breast cancer
* Prior biopsy exhibiting atypical hyperplasia or lobular carcinoma in situ (LCIS)
* History of invasive breast cancer or ductal carcinoma in situ (DCIS) and have completed standard therapy including tamoxifen/aromatase inhibitor or will not be treated with tamoxifen/aromatase inhibitor
* Signed Informed Consent

Exclusion Criteria:

* Metastatic breast cancer
* Undergoing treatment (chemotherapy, radiation, or SERMs)
* Pregnancy or breast-feeding, or planning to become pregnant within one year prior to study entry
* Regular soy consumers (i.e., < once per week of soy food, soy supplements or other products)
* Known food allergies such as to soy or nuts
* Not willing to avoid soy foods/supplements during study period
* Current users of exogenous hormones or oral contraceptive or planning to use exogenous hormones during the duration of the study
* Cannot stop taking aspirin or NSAIDs within a week of breast biopsy
* Active participant in other ongoing trials

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with reduced MRI volume (MRIV) | At completion of 12 months on the study

SECONDARY OUTCOMES:
Percentage of cells that stain positive for Ki67, caspase 3, ratio of Ki67/caspase, ER alpha and ER beta | At completion of 12 months on the study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wu, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Wu AH, Spicer D, Garcia A, Tseng CC, Hovanessian-Larsen L, Sheth P, Martin SE, Hawes D, Russell C, MacDonald H, Tripathy D, Su MY, Ursin G, Pike MC. Double-Blind Randomized 12-Month Soy Intervention Had No Effects on Breast MRI Fibroglandular Tissue Density or Mammographic Density. Cancer Prev Res (Phila). 2015 Oct;8(10):942-51. doi: 10.1158/1940-6207.CAPR-15-0125. Epub 2015 Aug 14. PMID 26276750